CLINICAL TRIAL: NCT02169427
Title: An Open-label Study in Healthy Male Subjects to Assess the Absorption, Distribution, Metabolism and Excretion of [14C]-Labelled BIA 9-1067 and Metabolites Following a Single Dose Oral Administration
Brief Title: An Open-label Study in Healthy Male Subjects to Assess the Absorption, Distribution, Metabolism and Excretion of [14C]-Labelled BIA 9-1067 and Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-122
Record Dates: First submitted 2012-01-24; First posted 2014-06-23 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); BIA 9-1067; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Opicapone (OPC) (Experimental): 100 mg OPC
  Interventions: Drug: OPC

INTERVENTIONS:
Drug: OPC — The drug substance of 100 mg OPC was administered as 1 capsule.
  Other Names: BIA 9-1067

SUMMARY:
The purpose of this study is to determine the rate and routes of excretion of OPC and the mass balance in urine, faeces and expired air.

DETAILED DESCRIPTION:
This was a single-centre, open-label ADME study in 6 healthy male subjects. Subjects received a single dose of 100 mg OPC, containing 3.39 MBq of [14C] OPC as oral capsules.

The study consisted of an eligibility screening period within 3 weeks prior to drug administration, admission on Day -1, a treatment period involving drug administration on Day 1 followed by matrix collections for PK purposes and safety evaluations up to Day 11, discharge on Day 11, six 24-hour hospitalizations on Days 14/15, 21/22 (+/ 1 day), 28/29 (+/- 1 day), 42/43 (+/- 2 days), 56/57 (+/- 2 days) and 77/78 (+/ 3 days) for PK sample collections, and a follow up visit performed at least 14 days after discharge from the last 24-hour hospitalization or at early discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male
2. Age: 18 - 55 years, inclusive
3. Body Mass Index (BMI): 18.0 - 30.0 kg/m2, inclusive Body weight (kg)and height2 (m2)
4. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks") and grapefruit (juice) from 48 hours prior to entry in the clinical research centre until discharge
5. Medical history without major pathology
6. Resting supine blood pressure and a resting pulse rate showing no clinically relevant deviations as judged by the MI
7. Computerised (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the MI
8. Willingness to use adequate contraception from the time of dosing until 3 months after the follow-up visit
9. All values for haematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the MI
10. Willingness to sign the written ICF

Exclusion Criteria:

1. Evidence of clinically relevant pathology
2. Mental handicap
3. History of relevant drug and/or food allergies
4. Regular/routine treatment with non-topical medications within 30 days prior to entrance into the clinical research centre
5. Smoking (less than 60 days prior to drug administration)
6. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
7. Use of concomitant medication, except for acetaminophen (paracetamol), which was allowed up to 3 days before entrance into the clinical research centre. Multivitamins and vitamin C were allowed up to 7 days before entrance into the clinical research centre. All other medication (including over the counter medication, health supplements, and herbal remedies such as St. John's wort extract) was to be stopped at least 14 days prior to entrance into the clinical research centre
8. Participation in a drug study within 60 days prior to drug administration. Participation in more than 3 other drug studies in the 10 months preceding administration of study drug
9. Donation of more than 50 mL of blood within 60 days prior to drug administration. Donation of more than 1.5 litres of blood in the 10 months preceding administration of study drug
10. Participation in another ADME study with a radiation burden -0.1 mSv in the period of 1 year before the start of the study
11. Exposure to radiation for diagnostic reasons (except dental X-rays and plain X rays of thorax and bony skeleton - excluding spinal column), during work or during participation in a medical study in the previous year
12. Irregular defecation pattern (less than once per 2 days)
13. Positive screen on drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol)
14. Intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
15. Positive screen on hepatitis B surface antigen (HBsAg)
16. Positive screen on anti-hepatitis C virus (HCV)
17. Positive screen on anti- human immunodeficiency virus (HIV) 1/2
18. Illness within 5 days prior to drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA, Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opicapone (OPC)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Opicapone (OPC)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Recovery of [14C]-Radioactivity
Description: AEurine: Cumulative Recovery of [14C]-Radioactivity in urine AEfaeces: Cumulative Recovery of [14C]-Radioactivity in urine AEair: Cumulative Recovery of [14C]-Radioactivity in urine AEtotal: Cumulative Recovery of [14C]-Radioactivity in urine
  Recovery % of dose has been derived from area under the excretion rate (to infinity) from 240h onwards
Time Frame: pre-dose and 0-6, 6-12, 12-24, 24-48, 48 72, 72-96, 96 120, 120-144, 144-168, 168-192, 192-216 and 216-240 hours post-dose; 24-hour collections on Days 14/15, 21/22, 28/29
Measure: Mean (Standard Deviation); unit: Recovery % of dose
Arm/Group | Opicapone (OPC)
Number analyzed (Participants) | 6
Recovery % of dose
  AEurine | 12.8 (1.5)
  AEfaeces | 67.2 (7.6)
  AEair | 15.9 (4.8)
  AEtotal | 95.9 (8.6)

2. Secondary Outcome: Cmax - Maximum Concentration
Description: BIA 9-1103 is a Opicapone (OPC, BIA 9-1067) metabolite
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng [eq]/mL
Arm/Group | Opicapone (OPC)
Number analyzed (Participants) | 6
ng [eq]/mL
  14C plasma | 7302 (3918)
  14C blood | 1920 (813)
  OPC plasma | 757 (321)
  BIA 9-1103 plasma | 118 (60.9)

3. Secondary Outcome: Tmax - Time to Attain Maximum Concentration
Description: BIA 9-1103 is a Opicapone (OPC, BIA 9-1067) metabolite
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Opicapone (OPC)
Number analyzed (Participants) | 6
hours
  14C plasma | 0.51 (0.01)
  14C blood | 1.01 (0.01)
  OPC plasma | 2.43 (1.10)
  BIA 9-1103 plasma | 8.34 (3.88)

ADVERSE EVENTS:
Arm/Group | Opicapone (OPC)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opicapone (OPC) (N=6)
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Wound (Injury, poisoning and procedural complications) | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other